CLINICAL TRIAL: NCT00468988
Title: Short Term Comparative Study of Xalatan With Benzalkonium Chloride vs. Travatan Z Without Benzalkonium Chloride in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SMA-06-21
Record Dates: First submitted 2007-05-02; First posted 2007-05-03 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Latanoprost

INTERVENTIONS:
Drug: Travatan® Z
Drug: Xalatan®

SUMMARY:
Compare the effect of Xalatan with benzalkonium chloride on the ocular surface to those effects observed with Travatan Z without benzalkonium chloride after a single dose

ELIGIBILITY:
Inclusion Criteria:

* Adults with primary open-angle glaucoma, ocular hypertension or pigment dispersion glaucoma

Exclusion Criteria:

* Age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-05; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Tear Break Up Time | Day

SECONDARY OUTCOMES:
Safety | Onset

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jasek, PhD, Study Director — Alcon Research
Locations (1):
- Orlando, Orlando, Florida, United States